CLINICAL TRIAL: NCT01623323
Title: A 3-Month Open-Label Multicenter Study Evaluating the Safety of Intranasal Administration of 400 μg of Fluticasone Propionate Twice a Day (BID) Using a Novel Bi-Directional Device in Subjects With Chronic Sinusitis With or Without Nasal Polyps
Brief Title: Study Evaluating the Safety of Intranasal Administration of 400 μg of Fluticasone Propionate Twice a Day (BID) Using a Novel Bi-Directional Device in Subjects With Chronic Sinusitis With or Without Nasal Polyps
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPN-FLU-CS-3204
Record Dates: First submitted 2012-06-14; First posted 2012-06-19 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Sinusitis With or Without Nasal Polyps
MeSH Terms: interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluticasone (Other)
  Interventions: Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Fluticasone Propionate — Fluticasone Propionate 400 μg

SUMMARY:
This is an open-label, multicenter study designed to assess the safety of intranasal administration of 400 μg of fluticasone propionate twice a day delivered by the OptiNose device in subjects with chronic sinusitis with or without nasal polyps. The study consists of an up-to-7-day pretreatment phase followed a 3-month open-label treatment phase. The duration of each subject's participation is approximately 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years and older
* Women must

  * be practicing an effective method of birth control (eg, prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method [eg, condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel], or male partner sterilization) before entry and throughout the study, or
  * be surgically sterile (have had a hysterectomy or bilateral oophorectomy, or tubal ligation at least 1 year before screening) or otherwise be incapable of pregnancy, or
  * be postmenopausal (spontaneous amenorrhea for at least 1 year).
* Women of child-bearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) pregnancy test at the screening visit
* Have either:

a history of chronic sinusitis with bilateral nasal polyposis determined by nasoendoscopy at screening visit OR a history of chronic sinusitis (without polyps) for equal to or greater than 12 weeks and currently experiencing 2 or more of the following symptoms, one of which MUST be either nasal blockage/congestion or nasal discharge (anterior and/or posterior nasal discharge):

1. nasal blockage/congestion
2. nasal discharge (anterior and/or posterior nasal discharge)
3. facial pain or pressure
4. reduction or loss of smell

   * Subjects with comorbid asthma or COPD must be stable with no exacerbations (eg, no emergency room visits, hospitalizations, or oral or parenteral steroid use) within the 3 months before the screening visit. Inhaled corticosteroid use must be limited to stable doses of no more than 1,000 μg/day of beclomethasone (or equivalent; See Attachment 1) for at least 3 months before screening with plans to continue use throughout the study.
   * Must be able to cease treatment with intranasal steroids and inhaled corticosteroids (except permitted doses listed above for asthma and COPD) at the screening visit
   * Must be able to use the OptiNose device correctly; all subjects will be required to demonstrate correct use of the placebo device at the screening visit, see Section 12.1, Visit 1, screening procedures.
   * Must be capable, in the opinion of the investigator, of providing informed consent to participate in the study. Subjects must sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Women who are pregnant or lactating
* Inability to have each nasal cavity examined for any reason, including nasal septum deviation
* Nasal septum perforation
* Has had more than 1 episode of epistaxis with frank bleeding in the month before the screening visit
* Have evidence of significant baseline mucosal injury, ulceration or erosion (eg, exposed cartilage, perforation) on baseline nasal examination/nasoendoscopy
* History of sinus or nasal surgery within 6 months before the screening visit
* Current, ongoing rhinitis medicamentosa (rebound rhinitis)
* Have significant oral structural abnormalities, eg, a cleft palate
* Diagnosis of cystic fibrosis
* History of Churg-Strauss syndrome or dyskinetic ciliary syndromes
* Purulent nasal infection, acute sinusitis, or upper respiratory tract infection within 2 weeks before the screening visit. Potential subjects presenting with any of these infections may be rescreened 4 weeks after symptom resolution
* Planned sinonasal surgery during the period of the study
* Allergy, hypersensitivity, or contraindication to corticosteroids or steroids
* Allergy or hypersensitivity to any excipients in study drug
* Exposure to any glucocorticoid treatment with potential for systemic effects (eg, oral, parenteral, intra-articular, or epidural steroids, high dose topical steroids) within 1 month before the screening visit; except as noted in inclusion criteria for subjects with comorbid asthma or COPD
* Have nasal candidiasis
* Have taken a potent CYP3A4 inhibitor within 14 days before the screening visit; examples of these medications can be found in Section 11.6, Concomitant Medication.
* History or current diagnosis of any form of glaucoma or ocular hypertension (ie, intraocular pressure >21 mmHg)
* History of intraocular pressure elevation on any form of steroid therapy
* History or current diagnosis of the presence (in either eye) of a cataract
* Any serious or unstable concurrent disease, psychiatric disorder, or any significant condition that, in the opinion of the investigator could confound the results of the study or could interfere with the subject's participation or compliance in the study
* A recent (within 1 year of the screening visit) clinically significant history of drug or alcohol use, abuse, or dependence that, in the opinion of the investigator could interfere with the subject's participation or compliance in the study
* Positive urine drug screen at screening visit for drugs of abuse (see Section 14.5), with the exception of prescribed medications for legitimate medical conditions
* Have participated in a previous clinical trial of OPTINOSE FLUTICASONE
* Have participated in an investigational drug clinical trial within 30 days of the screening visit
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Precision Trials, Phoenix, Arizona
  - Colorado ENT and Allergy, Colorado Springs, Colorado
  - Sher Allergy, Largo, Florida
  - ENT of Georgia, Decatur, Georgia
  - Best Clinical Trials, New Orleans, Louisiana
  - Institute for Asthma and Allergy, Wheaton, Maryland
  - Clinical Research Group of Montana, Bozeman, Montana
  - ENT and Allergy Associates, New Windsor, New York
  - ENT and Allergy Associates, West Nyack, New York
  - Vital Prospects Clinical Research Institute, Tulsa, Oklahoma
  - Allergy Associates Research Center, Portland, Oregon
  - Live Oak Allergy and Asthma Clinic, Live Oak, Texas
  - Texas Quest Medical Research, San Antonio, Texas
  - Focus Clinical Research, Draper, Utah
  - InterMountain Ear Nose and Throat, Salt Lake City, Utah
  - Chrysalis Clinical Research, St. George, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Premier Clinical Research, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- OPN-375: OPN-375 400 mcg/twice daily
Period: Overall Study
Arm/Group | OPN-375
Started | 705
Completed | 601
Not Completed | 104

BASELINE CHARACTERISTICS:
Arm/Group | OPN-375
Number analyzed (Participants) | 705
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (13.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 403
  Male | 302
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 81
  Not Hispanic or Latino | 624
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 28
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 114
  White | 552
  More than one race | 6
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 705

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Adverse Events were collected via spontaneous subject report and through physician examination. The display of adverse events is by subject.
Time Frame: Baseline to 3 months or End of Study
Population: All subject who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | OPN-375
Number analyzed (Participants) | 705
participants | 270

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | OPN-375
Serious Adverse Events (participants affected / at risk) | 5/705
Other Adverse Events (participants affected / at risk) | 180/705
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPN-375 (N=705)
acute cholecystitis (Hepatobiliary disorders) | 1 (1)
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPN-375 (N=705)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 102
Nasal Mucosal Disorder (Respiratory, thoracic and mediastinal disorders) | 72
Nasal Septal Disorder (Respiratory, thoracic and mediastinal disorders) | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days